CLINICAL TRIAL: NCT05249283
Title: Self and Body Perception in Otoneurological Disorders: Translation and Validation of Measurement Scales
Acronym: PERSOCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21-44
Record Dates: First submitted 2022-01-18; First posted 2022-02-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Patients With Acute or Chronic Otoneurological Disorders; Patients Presenting or Having Experienced Dizziness and / or Balance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Patients with acute or chronic otoneurological disorders, presenting or having experienced dizziness and / or balance disorders
  Interventions: Other: Questionnaire Measures
- Control subjects (Other)
  Interventions: Other: Questionnaire Measures

INTERVENTIONS:
Other: Questionnaire Measures — Patients will complete the following questionnaires: CDS questionnaire, Niigata PPPD questionnaire, HAD (Hospital Anxiety and Depression) scale and DHI (Dizziness Handicap Inventory)

SUMMARY:
Depersonalization-derealization (DD) disorders are a clinical phenomenon characterized by feeling disconnected or detached from one's self. Individuals may report feeling as if they are an outside observer of their own thoughts or body, and often report feeling a loss of control over their thoughts or actions.

Several scales have been developed to measure DD, and the Cambridge Depersonalization Scale (CDS) appears to be the most relevant and consistent to characterize the clinical symptoms of these disorders as well as their duration and frequency. This scale, originally written in English, must be translated and validated according to standardized methods that include testing steps patients with dizziness and in individuals with no vestibular disorder.

Persistent postural-perceptual dizziness (PPPD) is a chronic, persistent vestibular syndrome generally preceded by acute vestibular disorders. The main symptoms are rotational dizziness, unsteadiness and / or non-rotating dizziness that are exacerbated by upright posture, walking, active or passive movement, and exposure to moving visual stimuli or complex visual patterns. To help diagnose this syndrome, a questionnaire was developed in Japan in 2019, the Niigata questionnaire, however no French version has yet been validated. Similarly, this scale needs to be validated in patient with PPPD and in control populations.

The main objective of this study is to validate the French translation of these two scales, the CDS questionnaire and the Niigata PPPD questionnaire, according to standard methods (forward translation, back translation, consensus).

ELIGIBILITY:
Inclusion Criteria:

For patient:

* Age ≥ 18 years
* Patient with acute or chronic otoneurological disorders
* Patient having or having experienced dizziness and / or balance disorders
* Patient with PPPD
* Fluency in French
* Having given free and informed written consent
* Being affiliated with or benefiting from social security

For control subjects:

* Age ≥ 18 years
* Fluency in French
* Having given free and informed written consent
* Being affiliated with or benefiting from social security.

Exclusion Criteria:

For patient:

-Past or present psychiatric and neurological disease (other than otoneurological or PPPD, as declared by the participant)

For control subjects:

-Past or present psychiatric and neurological disease (as declared by the participant) and vestibular and/or auditory system disorders (as declared by the participant)

For all participants:

* Persons still in a period of exclusion from another study and persons simultaneously participating in another study
* Subject to a measure for the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Scores from the CDS questionnaire translated according to standardized methods (forward translation, back translation, consensus) in patients with other vestibular disorders and control subjects. | 24 months
Scores from the Niigata PPPD questionnaire translated according to standardized methods (forward translation, back translation, consensus) in patients with PPPD, patients with other vestibular disorders and control subjects. | 24 months

SECONDARY OUTCOMES:
Measurement of the HADS score in patients with PPPD, in patients with other vestibular disorders and in control subjects | 24 months
Measurement of the DHI score in patients with PPPD, patients with other vestibular disorders and control subjects | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No